CLINICAL TRIAL: NCT02084563
Title: Evaluation of the Incidence and Prognostic Impact of Molecular and Genetic Abnormalities in Patients With Acute Myeloid Leukemia, Myelodysplastic Syndrome and Myeloproliferative Neoplasms
Brief Title: Study of Molecular and Genetic Abnormalities in Patients With Myeloid Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Fabio Pires de Souza Santos, MD, Hospital Israelita Albert Einstein
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LMA Brasil; 11/1714 (Other: HIAE CEP)
Record Dates: First submitted 2013-01-02; First posted 2014-03-12 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Acute Myeloid Leukemia; Myeloproliferative Neoplasms; Myelodysplastic Syndromes; Myeloproliferative/Myelodysplastic Neoplasm
Keywords: Acute Myeloid Leukemia; Myeloproliferative Neoplasms; Myelodysplastic Syndromes; Myeloproliferative/Myelodysplastic Neoplasm; Leukemia; MDS; MPN; AML; Chronic myelomonocytic leukemia (CMML); Polycythemia Vera (PV); Essential Thrombocythemia (ET); Myelofibrosis (MF)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia; Leukemia, Myelomonocytic, Chronic; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — Induction Chemotherapy; Cytarabine; Daunorubicin; Anthracyclines; Consolidation Chemotherapy; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AML-Intensive Chemotherapy (Other): Patients with Acute Myeloid Leukemia fit for intensive chemotherapy Patients will receive Induction Chemotherapy, and CR will be evaluated after 28 days.
  Patients who achieve CR post-induction chemotherapy will receive post-remission therapy according to risk:
  * Low risk patients: Consolidation chemotherapy or Autologous stem cell transplantation
  * Intermediate and high-risk patients: Allogeneic stem cell transplantation Patients who do not achieve CR may receive one second induction cycle, and if CR is achieved may proceed to post-remission therapy as per above. Patients who do not achieve CR after two cycles of induction will be deemed refractory and removed from the study.
  Interventions: Drug: Induction Chemotherapy; Drug: Consolidation Chemotherapy; Drug: Autologous Stem Cell Transplantation; Drug: Allogeneic Stem Cell Transplantation
- AML-Non-intensive chemotherapy (Other): Patients with acute myeloid leukemia not fit for intensive chemotherapy Patients will receive induction chemotherapy with either low dose cytarabine or decitabine. Assignment to each drug will depend on drug availability and physician discretion. No randomization will be done between the drugs.
  Cycles will be repeated every 28 days. Patients who achieve CR will continue to post-consolidation therapy with either cytarabine or decitabine, based on the induction therapy received. Patients will receive a maximum of 4 cycles until achieving CR, if no response is seen after 4 cycles patients will be deemed refractory.
  Interventions: Drug: Low Dose Cytarabine; Drug: Decitabine
- Chronic Myeloid Disorders (No Intervention): Patients with Chronic Myeloid Disorders:
  * Myeloproliferative Neoplasms
  * Myelodysplastic Syndromes
  * Myeloproliferative/Myelodysplastic Neoplasms

INTERVENTIONS:
Drug: Induction Chemotherapy — Induction chemotherapy for patients with AML eligible for intensive chemotherapy:
  * Cytarabine 200 mg/m2 IV continuous infusion days 1-7
  * Daunorubicin 90 mg/m2 intravenous piggyback days 1-3
  Other Names: 7+3; Ara-C; Daunorubicin; Anthracycline; 3+7
  Arms: AML-Intensive Chemotherapy
Drug: Consolidation Chemotherapy — Consolidation chemotherapy for patients eligible for intensive chemotherapy with low-risk AML or patients with intermediate-/high-risk AML who do not have matched donors:
  -Cytarabine 1.5 g/m2 IV in 3 hours days 1, 3 and 5 for 3 cycles
  Other Names: Ara-C; Cytarabine
  Arms: AML-Intensive Chemotherapy
Drug: Autologous Stem Cell Transplantation — Autologous Stem Cell Transplantation for consolidation of patients eligible for intensive chemotherapy with low-risk AML or patients with intermediate-/high-risk AML who do not have matched donors:
  * Busulfan 1 mg/Kg PO q6h or 130 mg/m2 IV once daily days -7 to -4
  * Cyclophosphamide 60 mg/Kg IV once daily days -3 and -2
  Other Names: ASCT; Autologous Bone Marrow Transplantation; ABMT
  Arms: AML-Intensive Chemotherapy
Drug: Allogeneic Stem Cell Transplantation — Allogeneic Stem Cell Transplantation for consolidation of patients eligible for intensive chemotherapy with intermediate-/high-risk AML
  Conditioning regimen:
  * Busulfan 1 mg/Kg PO q6h or 130 mg/m2 IV once daily days -7 to -4
  * Cyclophosphamide 60 mg/Kg IV once daily days -3 and -2 or Fludarabine 40 mg/m2 IV once daily days -7 to -4
  Other Names: AlloSCT; Allogeneic Bone Marrow Transplantation
  Arms: AML-Intensive Chemotherapy
Drug: Low Dose Cytarabine — Chemotherapy for patients with AML who are not fit for intensive chemotherapy:
  * Cytarabine 60 mg/m2 subcutaneous (SQ) bid days 1-5 (until CR or maximum 4 cycles)
  * Cytarabine 40 mg/m2 SQ bid days 1-5 (after CR, until a maximum of 3 years of therapy or relapse, whichever comes first)
  Other Names: Low dose ara-C; LDAC
  Arms: AML-Non-intensive chemotherapy
Drug: Decitabine — Chemotherapy for patients with AML who are not fit for intensive chemotherapy:
  * Decitabine 20 mg/m2 IV once daily days 1-10 (until CR or maximum 4 cycles)
  * Decitabine 20 mg/m2 IV once daily days 1-5 (after CR, until a maximum of 3 years of therapy or relapse, whichever comes first)
  Other Names: 2-aza-5´-deoxycytidine; Dacogen; DAC
  Arms: AML-Non-intensive chemotherapy

SUMMARY:
The objective of this study is to describe the prevalence and prognostic impact of the most common genetic abnormalities in patients with Myeloid Neoplasms, including Acute Myeloid Leukemia (AML), Myeloproliferative Neoplasms (MPN), Myelodysplastic Syndromes (MDS) and Myeloproliferative/Myelodysplastic Neoplasms. Patients will have samples of blood and/or bone marrow collected and sent to Hospital Israelita Albert Einstein for analysis and storage.

Patients with a diagnosis of Acute Myeloid Leukemia will be treated according to an uniform protocol.

ELIGIBILITY:
Acute Myeloid Leukemia-Intensive Chemotherapy

Inclusion Criteria:

* Diagnosis of AML according to WHO criteria
* Age greater than 18 years
* Performance status (ECOG) between 0-2
* Adequate liver and kidney function
* Signed Informed Consent form
* No prior therapy for AML, except use of hydroxyurea for control of elevated white blood cell counts
* Adequate contraception for fertile men and women
* Eligible for intensive chemotherapy (as judged by the treating physician)

Exclusion Criteria:

* Acute myeloid leukemia with retinoic acid receptor alpha (RARA) translocations (APL, acute promyelocytic leukemia)
* Pregnant women
* HIV-positivity
* New York Heart Association class III and IV congestive heart failure
* Patient refuses to use adequate contraception
* History of hypersensibility to any of the used chemotherapy drugs
* Patient refuses to sign informed consent form

Acute Myeloid Leukemia-Non-Intensive Chemotherapy

Inclusion Criteria:

* Diagnosis of AML according to WHO criteria
* Age greater than 18 years
* Signed Informed Consent form
* No prior therapy for AML, except use of hydroxyurea for control of elevated white blood cell counts
* Adequate contraception for fertile men and women
* Non-eligible for intensive chemotherapy (as judged by the treating physician)

Exclusion Criteria:

* Acute myeloid leukemia with RARA translocations (APL, acute promyelocytic leukemia)
* Pregnant women
* HIV-positivity
* Patient refuses to use adequate contraception
* History of hypersensibility to any of the used chemotherapy drugs
* Patient refuses to sign informed consent form

Chronic Myeloid Disorders:

Inclusion Criteria:

* Diagnosis of Myeloproliferative Neoplasm or Myelodysplastic Syndrome or Myeloproliferative/Myelodysplastic Neoplasm according to WHO criteria
* Age greater than 18 years
* Signed Informed Consent form

Exclusion Criteria:

* Patient refuses to sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of molecular and cytogenetic abnormalities | 2 years
  As assessed by results of molecular and cytogenetic tests and frequency in the population studied

SECONDARY OUTCOMES:
Overall survival | 5 years
  Evaluation of 5-years overall survival in patients with Acute Myeloid Leukemia, Myeloproliferative Neoplasms, Myelodysplastic Syndromes and Myeloproliferative/Myelodysplastic Neoplasms
Response rate | 1 month
  Evaluate complete remission (CR) rate at 1 month for patients with Acute Myeloid Leukemia who received induction chemotherapy. Complete remission was defined by the presence of < 5% blasts in the bone marrow (BM) with > 1 x 10^9/L neutrophils and >100x10^9/L platelets in the peripheral blood (PB)
Disease Free Survival | 5 years
  Evaluate rate of 5-years disease-free survival in patients with Acute Myeloid Leukemia who enter complete remission after induction chemotherapy
Cumulative incidence of relapse and non-relapse mortality | 5 years
  Evaluate 5-years cumulative incidence of relapse and non-relapse mortality in patients with Acute Myeloid Leukemia who achieve complete remission following induction chemotherapy
Number of participants with adverse events as a measure of safety and tolerability | 1 year
  Evaluate hematological and non-hematological toxicity in patients with Acute Myeloid Leukemia treated according to the protocol. Toxicity will be graded as per the National Cancer Institute Common Toxicity Criteria for Adverse Events v4.0.3
Cumulative Incidence of Transformation to Acute Myeloid Leukemia | 5 years
  Evaluate 5-years incidence of transformation to Acute Myeloid Leukemia in patients with Myeloproliferative Neoplasms, Myelodysplastic Syndromes and Myeloproliferative/Myelodysplastic Neoplasms

CONTACTS AND LOCATIONS:
Overall Officials: Fabio P Santos, MD, Study Director — Hospital Israelita Albert Einstein; Nelson Hamerschlak, MD, PhD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil